CLINICAL TRIAL: NCT06827678
Title: Establishment of the Chinese Preclinical Alzheimer's Disease Study With Multiple Neuroimaging
Status: Recruiting | Type: Observational
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, YiHui Guan, Professor, Huashan Hospital
Other Study IDs: KY2024-723
Record Dates: First submitted 2024-12-05; First posted 2025-02-14 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease; Positron Emission Tomography
Keywords: Alzheimer's Disease; PET imaging; Biomarker; Body Imaging
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from Blood will be collected

GROUPS / COHORTS (1):
- Chinese Preclinical Alzheimer's Disease Study: This cohort will included AD, MCI and Cognitively un-impairments.
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No intervention

SUMMARY:
The goal of this observational study is to investigate neuroimage and biomarkers in the Alzheimer's continuum in Chinese population. We aimed to:

* To reveal the progress of AD by multiple neuroimage and biomarkers;
* To reveal the longitudinal change of biomarkers and cognition of AD in Chinese population;
* To investigate the interaction of markers between body and brain;
* To set up new markers by neuroimage.

DETAILED DESCRIPTION:
The observational study is recruiting participants from clinics and communities with cognitive impairments and un-impairments. As the part of our previous study: Chinese Preclinical Alzheimer's Disease Study (C-PAS) cohort. We will include lager size of body and brain PET imaging. The study will also integrate multi-dimensional scales, peripheral biomarkers, metabolites, electroencephalograms, genetics, and other indicators for multi-omics analysis to deeply explore the mechanisms underlying the onset and progression of Alzheimer's disease. By identifying risk factors closely associated with Alzheimer's disease, we aim to develop a comprehensive disease risk model, providing reliable evidence for early detection and prevention, and uncovering new targets for therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Cognitive unimpaired(CU) controls:

(1) Aged between 45 and 90 years; no gender restrictions； (2) Cognitive function is assessed as normal by the researcher based on cognitive tests, with a Clinical Dementia Rating (CDR) score of 0; (3) Confirmed by the researcher to have no neurological diseases, major chronic illnesses, malignant tumors, or acute infectious diseases; (4) No family history of Alzheimer's disease (AD) or other neurological diseases related to cognitive impairment and movement disorders; (5) Able to understand and provide written informed consent before any assessment; (6) Female subjects must provide medical documentation proving they have undergone surgical sterilization (e.g., hysterectomy, bilateral oophorectomy, or tubal ligation) or have been menopausal for over one year. If they are still of childbearing potential, they must use effective contraceptive measures during the study; (7) Male subjects must use effective contraceptive measures during the study period and are prohibited from donating sperm during this time; (8) Willing and able to comply with all study procedures. 2. Cognitive impaired(CI) patients:

1. Aged between 45 and 90 years; no gender restrictions;
2. CDR score ≥ 0.5;
3. MMSE score ≤ 24;
4. Brain MRI findings support the diagnosis of AD, with no evidence of other neurological diseases;
5. Any medications taken to alleviate AD symptoms must be maintained at a stable dose for at least 30 days before study participation;
6. Written informed consent must be provided by the subject or their legal guardian/caregiver;
7. If necessary, subjects may be accompanied by a caregiver;
8. Before any assessment, the subject or their legal representative must understand and sign a written informed consent form;
9. Female subjects must provide medical documentation confirming surgical sterilization (e.g., hysterectomy, bilateral oophorectomy, or tubal ligation).

Exclusion Criteria:

* All subjects:

  1. Presence of severe neurological diseases or serious disorders affecting the gastrointestinal, cardiovascular, hepatic, renal, hematologic, oncologic, endocrine, respiratory, or immune systems;
  2. Presence of MRI-incompatible metal implants, including cardiac pacemakers, intravascular metal devices, insulin pumps, cochlear implants, nerve stimulators, or cerebral aneurysm clips;
  3. Inability to tolerate MRI noise or a history of claustrophobia;
  4. Exposure to ionizing radiation exceeding 50 mSv within the past year due to participation in other clinical or scientific research;
  5. History of drug or alcohol abuse;
  6. Pregnancy or lactation;
  7. Poor venous access, making repeated venipuncture infeasible;
  8. Use of experimental drugs or devices with unknown efficacy or safety within the past month;
  9. Allergy to any components of the tracer injection;
  10. Any condition that, in the investigator's judgment, may pose a risk or compromise the integrity of the study.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are recruited from neurology outpatient clinics and community settings.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Synaptic Density in Alzheimer's Disease Using Synaptic Vesicle Glycoprotein 2A (SV2A) PET Tracer [¹⁸F]SDM-8 | 90 minutes post-injection
  Subjects received an intravenous injection of the radiopharmaceutical at a dose of 1.8 MBq/kg (0.05 mCi/kg). After a 90-minute rest in a quiet, light-controlled room, PET imaging was performed using a PET/CT or PET/MRI scanner with a dedicated head protocol. Scanning was conducted in 3D mode (FOV: 180 mm), and images were reconstructed using the 3D RAMLA algorithm at a resolution of 2×2×2 mm. PET images were co-registered with structural CT or MRI scans. For quantitative analysis, target regions, including cortical areas and the cerebellum, were delineated on normalized structural images and projected onto PET images to measure radiotracer uptake. The standardized uptake value ratio (SUVr) was calculated as the ratio of cortical to cerebellar uptake.
Evaluation of Neuronal Function in Alzheimer's Disease Using Metabotropic Glutamate Receptor 5 (mGluR5) PET Tracer [¹⁸F]PS232 | 90 minutes post-injection
  Subjects received an intravenous injection of the radiopharmaceutical at a dose of 1.8 MBq/kg (0.05 mCi/kg). After a 90-minute rest in a quiet, light-controlled room, PET imaging was performed using a PET/CT or PET/MRI scanner with a dedicated head protocol. Scanning was conducted in 3D mode (FOV: 180 mm), and images were reconstructed using the 3D RAMLA algorithm at a resolution of 2×2×2 mm. PET images were co-registered with structural CT or MRI scans. For quantitative analysis, target regions, including cortical areas and the cerebellum, were delineated on normalized structural images and projected onto PET images to measure radiotracer uptake. The standardized uptake value ratio (SUVr) was calculated as the ratio of cortical to cerebellar uptake.

SECONDARY OUTCOMES:
Multi-sequence MR Imaging Data Collection | A 5-year follow-up with assessments conducted annually.
  This multi-sequence MRI approach allows for the early detection of neurodegenerative changes, tracking of synaptic and vascular alterations, and identification of atrophy patterns associated with cognitive decline. Each subject underwent MRI scanning using a Siemens Prisma 3.0T research MRI scanner. The acquisition sequences included T1WI, T2WI, DTI, ASL, SWI, and rs-fMRI, which provide comprehensive structural, functional, and perfusion-related information on brain integrity. These sequences were also collected during follow-up assessments.
Peripheral Blood Biomarker Collection | A 5-year follow-up with assessments conducted annually.
  Blood-based biomarkers offer a minimally invasive method for detecting Alzheimer's disease-related pathology and monitoring disease progression , including tau pathology, neuroinflammation, and glial activation. Peripheral blood biomarker data, including p-tau181, p-tau231, p-tau217, GFAP, sTREM2, etc., were collected to assess neurodegeneration and neuroinflammation. Plasma samples were stored at -80 °C and analyzed using the Quanterix Simoa HD-1 platform. Measurements were conducted by technicians blinded to clinical imaging data. The concentrations of these plasma biomarkers are presented in pg/mL.
Neuropsychological Scale Assessment | A 5-year follow-up with assessments conducted annually.
  Neuropsychological assessments provide crucial insights into cognitive decline, aiding in the early diagnosis of Alzheimer's disease and other dementias. Cognitive function was assessed using standardized neuropsychological scales, including MMSE (minimum value 0, maximum value 30, higher scores indicate better cognitive function) and MoCA-B (minimum value 0, maximum value 30, higher scores indicate better cognitive function), among others.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Xie, PhD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided